CLINICAL TRIAL: NCT02559024
Title: Phase I/Ib Study of Surgical Resection or Radiofrequency Ablation (RFA) of Metastatic Lesions in the Liver in Combination With Monoclonal Antibody to OX40 (MEDI6469) in Patients With Metastatic Colorectal Cancer
Brief Title: Anti-OX40 Antibody (MEDI6469) in Patients With Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug expired and access to additional supply ended. PI left the institution shortly afterwards and the study will not be re-activated. Only 4 patients were enrolled.
Sponsor: Providence Health & Services (Other)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-102A
Record Dates: First submitted 2015-09-22; First posted 2015-09-24 (Estimated); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Colorectal Neoplasms
Keywords: Metastatic colorectal cancer; liver lesion; anti-OX40 antibody; MEDI6469; Immunotherapy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 21 Days (Experimental): MEDI6469 0.4 mg/kg IV x 3 doses over 5-6 days starting 21 days prior to surgery
  Interventions: Drug: MEDI6469
- 14 Days (Experimental): MEDI6469 0.4 mg/kg IV x 3 doses over 5-6 days starting 14 days prior to surgery
  Interventions: Drug: MEDI6469
- 7 Days (Experimental): MEDI6469 0.4 mg/kg IV x 3 doses over 5-6 days starting 7 days prior to surgery
  Interventions: Drug: MEDI6469

INTERVENTIONS:
Drug: MEDI6469 — MEDI6469 0.4 mg/kg IV x 3 doses over 5-6 days
  Other Names: anti-OX40 antibody; CD134

SUMMARY:
This study will test the ability of an immune modulator, anti-OX40 (MEDI6469) to alter the immune cell environment within colorectal cancer metastases. The drug will be administered to patients before surgical treatment.

DETAILED DESCRIPTION:
There will be three distinct cohorts of patients which will vary the timing of the MEDI6469 dose, starting three weeks before surgery and decreasing the interval before surgery by one week with each cohort, as long as no dose-limiting toxicity attributable to the anti-OX40 are observed.

Immunohistochemistry will be used to measure the immune cells within primary and metastatic tumors when resected tissue is available, and surgically ablated tumors, giving each specimen an "immune score". The primary endpoint of the study will be the difference in immune scores of patients treated with anti-OX40 compared to historical controls (immune scores of untreated patients). Secondary endpoints will include both clinical (survival) and immunological data (specific measurements of immune cell populations based on flow cytometry and immunohistochemistry).

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo staged liver resections are included in this study. In these cases, preoperative MEDI6469 will be given prior to the initial procedure.
* Patients with small <3 cm tumors located >2 cm away from central bile ducts will be considered for either radiofrequency ablation or resection, the choice of which will be determined at the time of surgery.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Laboratory values during preoperative assessment within the protocol specified range
* Ability to give informed consent and comply with the protocol. Patients with a history of psychiatric illness must be judged able to understand the investigational nature of the study and the risks associated with the therapy.
* No active gastrointestinal bleeding.
* No clinical or laboratory coagulopathy
* Anticipated lifespan greater than 12 weeks

Exclusion Criteria:

* Metastatic disease outside of the liver that is not considered surgically resectable or curable.
* Active infection.
* Active autoimmune disease including patients with Inflammatory Bowel Disease as determined by an autoimmune questionnaire.
* Previous treatment with mouse monoclonal antibodies.
* Need for chronic maintenance oral steroids.
* Any medical or psychiatric condition that in the opinion of the PI would preclude compliance with study procedures.
* Enrollment in a clinical trial in which a different investigational agent is administered within 4 weeks prior to the first dose of MEDI6469.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-03-14 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Safety (side-effects or complications related to the study drug) | 48 Days
  Patients are seen at least 7 times in clinic and have 3 physical exams and provide interim medical history four times to identify potential side-effects or complications related to the study drug.
Immune Score | 27 Days
  The number of CD8 effector T cells, CD4 regulatory T cells, the expression of activation markers OX40, CD38 and HLA-DR.

CONTACTS AND LOCATIONS:
Overall Officials: Pippa Newell, MD, Principal Investigator — Providence Health & Services
Locations (1):
- Portland Providence Medical Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Providence Cancer Center — http://oregon.providence.org/our-services/p/providence-cancer-center/